CLINICAL TRIAL: NCT02260180
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of the Dose-Response Profile of A-101 Topical Solution in Subjects With Seborrheic Keratosis of the Face
Brief Title: Study of A-101 for the Treatment of Seborrheic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-203
Record Dates: First submitted 2014-10-03; First posted 2014-10-09 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A-101 40% (Active Comparator): A-101 40% Topical Solution
  Interventions: Drug: A-101
- A-101 32.5% (Active Comparator): A-101 32.5% Topical Solution
  Interventions: Drug: A-101
- A-101 Vehicle Topical Solution (Placebo Comparator): A-101 0% Topical Solution (vehicle)
  Interventions: Drug: A-101

INTERVENTIONS:
Drug: A-101 — Topical Solution

SUMMARY:
The purpose of this study is to evaluate the safety and dose-response of 2 concentrations of A-101 versus a vehicle control in the treatment of seborrheic keratosis.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the dose-response relationship of 2 concentrations of A-101 Solution and its matching A-101 Solution Vehicle when applied to seborrheic Keratosis (SK) target lesions on the face. A further objective is to evaluate the safety and efficacy of 2 concentrations of A-101 Solution and its matching A-101 Solution Vehicle when applied topically up to 2 times to SK target lesions on the face.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject has a Fitzpatrick skin type of 1-4
3. Subject has a clinical diagnosis of stable clinically typical seborrheic keratosis
4. Subject has 1 appropriate seborrheic keratosis target lesion, as defined below (Section 5.4), on the face:

   * Have a clinically typical appearance
   * Be treatment naïve
   * Have a Physician's Lesion Assessment (PLA) of ≥2 (Section 6.1.2)
   * Have a longest axis that is ≥7mm and ≤15mm (Section 5.4)
   * Have a longest dimension perpendicular to the longest axis that is ≥7mm and ≤15mm (Section 5.4)
   * Have a thickness that is ≤2mm
   * Be a discrete lesion
   * Be, when centered in the area outlined by the provided 3cm diameter circular template, the only seborrheic keratosis lesion present
   * Not be on the eyelids
   * Not be within 5mm of the orbital rim
   * Not be covered with hair which, in the investigator's opinion, would interfere with the study medication application or the study evaluations (NB: the study medication may bleach hair)
   * Not be in an intertriginous fold
   * Not be pedunculated.
5. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an approved effective method of birth control (Section 8) for the duration of the study
6. Subject is non-pregnant and non-lactating
7. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of the target lesion or which exposes the subject to an unacceptable risk by study participation
8. Subject is willing and able to follow all study instructions and to attend all study visits
9. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Subject has clinically atypical and/or rapidly growing seborrheic keratosis lesions
2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Leser-Trelat)
3. Subject has a current systemic malignancy
4. Subject has a history of keloid formation or hypertrophic scarring
5. Subject has used any of the following systemic therapies within the specified period prior to Visit 1:

   * Retinoids; 180 days
   * Glucocortico-steroids; 28 days
   * Anti-metabolites (e.g., methotrexate); 28 days
6. Subject has used any of the following topical therapies within the specified period prior to Visit 1 on, or in a proximity to the target lesion, which in the investigator's opinion, interferes with the application of the study medication or the study assessments:

   * LASER, light (e.g., intense pulsed light (IPL), photo-dynamic therapy(PDT)) or other energy based therapy; 180 days
   * Retinoids; 28 days
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 60 days
   * Glucocortico-steroids or antibiotics; 14 days
7. Subject currently has or has had any of the following within the specified period prior to Visit 1 on, or in a proximity to the target lesion, which in the investigator's opinion, interferes with the application of the study medication or the study assessments :

   * A cutaneous malignancy; 180 days
   * Experienced a sunburn; 28 days
   * A pre-malignancy (e.g., actinic keratosis); currently
   * Body art (e.g., tattoos, piercing, etc.); currently
   * Excessive tan; currently
8. Subject has a history of sensitivity to any of the ingredients in the study medications
9. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, excessive hair, open wounds) which, in the investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
10. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Beger, BS, Study Director — Aclaris Therapeutics, Inc.
Locations (4):
- United States (4):
  - Oregon Medical Research Center, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - DermReseach, Inc., Austin, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 40% Topical Solution: A-101 40% Topical Solution
  A-101: Topical Solution
- A-101 32.5% Topical Solution: A-101 32.5% Topical Solution
  A-101: Topical Solution
Period: Overall Study
Arm/Group | A-101 40% Topical Solution | A-101 32.5% Topical Solution | A-101 Vehicle Topical Solution
Started | 39 | 39 | 41
Completed | 37 | 39 | 40
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-101 40% | A-101 32.5% | A-101 Vehicle Topical Solution | Total
Number analyzed (Participants) | 39 | 39 | 41 | 119
Age, Customized [Mean (Full Range); unit: years]
  Age | 71 [53 to 93] | 71 [33 to 88] | 67 [47 to 87] | 70 [33 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 20 | 65
  Male | 18 | 15 | 21 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 38 | 39 | 41 | 118
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of PLA Responders With Target Lesion Clear (PLA = 0) in Each Arm at Visit 8.
Description: The primary effectiveness analysis was a comparison between each A-101 group and the vehicle group based on the percentage with target lesions judged to be clear on the PLA (PLA = 0) at Visit 8. The three arms of the study are A-101 40% Topical Solution, A-101 32.5% Topical Solution, and A-101 0% Topical Solution (vehicle). The Physician's Lesion Analysis ( PLA) is a 4 point scale from 0 to 3, with 0 being lesion clear and 3 being the most severe lesion. A larger proportion of subjects with a PLA =0 is better.
Time Frame: Day 106
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 40% | A-101 32.5% | A-101 Vehicle Topical Solution
Number analyzed (Participants) | 37 | 39 | 40
Participants | 22 | 18 | 1
Statistical Analysis 1: Comparison: A-101 40% vs A-101 Vehicle Topical Solution; Test type: Superiority — 2-tail alpha was set to 0.05 with no adjustment for multiple comparisons; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: A-101 32.5% vs A-101 Vehicle Topical Solution; Test type: Superiority; p < 0.0001, Chi-squared; 2-tail alpha was set to 0.05 with no adjustment for multiple comparisons

2. Secondary Outcome: Mean Change From Baseline PLA Score at Visit 8
Description: A secondary efficacy analysis was the mean change from baseline PLA Score at visit 8. The three arms of the study are A-101 40% Topical Solution, A-101 32.5% Topical Solution, and A-101 0% Topical Solution (vehicle). The Physician's Lesion Analysis ( PLA) is a 4 point scale from 0 to 3, with 0 being lesion clear and 3 being the most severe lesion. A larger proportion of subjects with a PLA =0 is better. A lower (more negative) mean change is a better outcome.
Time Frame: Day 106
Population: Participants completing the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-101 40% | A-101 32.5% | A-101 Vehicle Topical Solution
Number analyzed (Participants) | 37 | 39 | 40
score on a scale | -1.7 (1.11) | -1.4 (1.14) | -0.1 (0.56)
Statistical Analysis 1: Comparison: A-101 40% vs A-101 Vehicle Topical Solution; Test type: Superiority; p < 0.0001, ANCOVA — No adjustment for multiple comparisons were made; Baseline PLA was the covariate. Comparisons were performed within the model using least-squares means and the common error term
Statistical Analysis 2: Comparison: A-101 32.5% vs A-101 Vehicle Topical Solution; The primary efficacy analysis of mean change from baseline to Visit 8 PLA was performed using analysis of covariance (ANCOVA) with baseline PLA as the covariate. Comparisons between vehicle and each A-101 group were performed within the model using least-squares means and the common error term; Test type: Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons were conducted; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) had a start date on or after the date of Visit 2 (study day 1) and treatment-emergent serious adverse events (TESAEs) had a start date on or after the date of Visit 1 (Screening). Collection continued through the patients last visit or the end of the study, visit 8 (Day 106.)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | A-101 40% | A-101 32.5% | A-101 Vehicle Topical Solution
All-Cause Mortality (participants affected / at risk) | 1/39 | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/39 | 0/39 | 1/41
Other Adverse Events (participants affected / at risk) | 13/39 | 7/39 | 12/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 40% (N=39) | A-101 32.5% (N=39) | A-101 Vehicle Topical Solution (N=41)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 40% (N=39) | A-101 32.5% (N=39) | A-101 Vehicle Topical Solution (N=41)
Eustacian Tube Obstruction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 3 (3) | 2 (2) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abcess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypocholestersterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02260180/Prot_SAP_000.pdf